CLINICAL TRIAL: NCT00115167
Title: A Multicenter, Randomised, Double-Blind, Placebo-Controlled Roll Over Study to Protocol 20010103 of Darbepoetin Alfa for the Treatment of Anemia of Cancer
Brief Title: A Study of Darbepoetin Alfa in Anemic Subjects Not Receiving Chemotherapy Who Have Completed the 20010103 Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20020149
Record Dates: First submitted 2005-06-21; First posted 2005-06-22 (Estimated); Last update posted 2009-05-11 (Estimated); Status verified 2009-05

CONDITIONS: Anemia; Cancer
Keywords: Oncology; Cancer-related anemia
MeSH Terms: conditions — Anemia; Neoplasms | interventions — Darbepoetin alfa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Darbepoetin alfa (Experimental)
  Interventions: Drug: Darbepoetin alfa
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Q4W
  Arms: Placebo
Drug: Darbepoetin alfa — Q4W
  Arms: Darbepoetin alfa

SUMMARY:
The purpose of this study is to determine the safety of darbepoetin alfa beyond 16 weeks of treatment in subjects with anemia of cancer who are not receiving chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

- Subjects completing the planned 16 weeks of treatment on the 20010103 Anemia of Cancer protocol

Exclusion Criteria:

* Subjects currently receiving or planned to receive cytotoxic chemotherapy or myelosuppressive radiotherapy
* Subjects who have other diagnoses not related to the cancer which can cause anemia
* Known history of seizure disorder
* Cardiac condition: uncontrolled angina, congestive heart failure, known ejection fraction less than 40%, or uncontrolled cardiac arrhythmia
* Uncontrolled hypertension
* Clinically significant systemic infection or chronic inflammatory disease present at the time of enrollment
* Subject of reproductive potential who is not using adequate contraceptive precautions
* Concerns for subject's compliance with the protocol procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 371 (Actual)
Dates: Start 2004-08; Primary Completion 2007-01 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | throughout study

SECONDARY OUTCOMES:
Confirmed antibody formation to investigational product | throughout study
Deaths on study | on study
Laboratory parameters | throughout study
Vital signs (blood pressure) | throughout study
Change in PRO scores | from baseline to end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Derived] Smith RE Jr, Aapro MS, Ludwig H, Pinter T, Smakal M, Ciuleanu TE, Chen L, Lillie T, Glaspy JA. Darbepoetin alpha for the treatment of anemia in patients with active cancer not receiving chemotherapy or radiotherapy: results of a phase III, multicenter, randomized, double-blind, placebo-controlled study. J Clin Oncol. 2008 Mar 1;26(7):1040-50. doi: 10.1200/JCO.2007.14.2885. Epub 2008 Jan 28. PMID 18227526
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com
- See also: Notice regarding posted summaries of trial results — http://download.veritasmedicine.com/REGFILES/amgen/Amgen_results_disclaimer.pdf
- See also: To access clinical trial results information click on this link — http://download.veritasmedicine.com/REGFILES/amgen/08D_FDAMA_113_Posting_Summary_33_NESP_20020149.pdf
- See also: FDA-approved Drug Labeling — http://www.aranesp.com/